CLINICAL TRIAL: NCT05959356
Title: Cetuximab and Envafolimab Plus mFOLFOXIRI Versus Cetuximab Plus mFOLFOX6 as First-line Treatment for RAS/BRAF Wild-type, MSS, Unresectable Left-side Metastatic Colorectal Cancer: A Randomized Controlled Phase II Trial (CEIL)
Brief Title: Cetuximab and Envafolimab Plus mFOLFOXIRI as First-line Treatment for RAS/BRAF Wild-type, MSS, Unresectable Left-side Metastatic Colorectal Cancer
Acronym: CEIL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU-33
Record Dates: First submitted 2023-07-16; First posted 2023-07-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: First-line treatment; RAS/BRAF wild-type; Microsatellite stable(MSS); Unresectable left-side metastatic colorectal cancer; Envafolimab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; envafolimab; Irinotecan; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): cetuximab+envafolimab+mFOLFOXIRI up to 8 cycles followed by maintenance with cetuximab+envafolimab+5-FU/LV
  Interventions: Drug: Cetuximab + Envafolimab + mFOLFOXIRI
- Arm B (Active Comparator): cetuximab+mFOLFOX6 up to 8 cycles followed by maintenance with cetuximab+5-FU/LV
  Interventions: Drug: Cetuximab + mFOLFOX6

INTERVENTIONS:
Drug: Cetuximab + Envafolimab + mFOLFOXIRI — Cetuximab 500mg/m² + envafolimab 200mg + irinotecan 150 mg/m² + oxaliplatin 85 mg/m² + leucovorin 200 mg/m² + 5-FU 2400 mg/m² civ. 46h all on day 1 of each 2 weeks cycle up to max 8 cycles, followed by maintenance with cetuximab 500mg/m² + envafolimab 200mg + leucovorin 200 mg/m² + 5-FU 400 mg/m² + 5-FU 2400 mg/m² civ. 46h all on day 1 of each 2 weeks cycle until PD, unacceptable toxicity or patient's refusal.
  Other Names: Cetuximab or c225; Envafolimab; Irinotecan; Oxaliplatin; Leucovorin; 5-FU
  Arms: Arm A
Drug: Cetuximab + mFOLFOX6 — Cetuximab 500mg/m² + oxaliplatin 85 mg/m² + leucovorin 200 mg/m² + 5-FU 400 mg/m² + 5-FU 2400 mg/m² civ. 46h all on day 1 of each 2 weeks cycle up to max 8 cycles, followed by maintenance with cetuximab 500mg/m² + leucovorin 200 mg/m² + 5-FU 400 mg/m² + 5-FU 2400 mg/m² civ. 46h all on day 1 of each 2 weeks cycle until PD, unacceptable toxicity or patient's refusal.
  Other Names: Cetuximab or c225; Oxaliplatin; Leucovorin; 5-FU
  Arms: Arm B

SUMMARY:
The primary aim of phase II CEIL study is to evaluate the efficacy of cetuximab and envafolimab plus mFOLFOXIRI versus cetuximab plus mFOLFOX6 as first line treatment of patients with initially unresectable and previously untreated RAS/BRAF wild-type, MSS, left-side metastatic colorectal cancer(mCRC), in terms of Progression-free Survival.

DETAILED DESCRIPTION:
This is a prospective, open-label, multi-center, randomized controlled phase II trial in which patients with initially unresectable and previously untreated RAS/BRAF wild-type, MSS, left-side mCRC will be randomized to two therapy groups:

Experimental arm A: receive induction treatment with cetuximab and envafolimab plus mFOLFOXIRI up to 8 cycles followed by maintenance with cetuximab and envafolimab plus 5-FU/LV until disease progression, unacceptable toxicity or patient's refusal.

Standard arm B: receive induction treatment with cetuximab plus mFOLFOX6 up to 8 cycles followed by maintenance with cetuximab plus 5-FU/LV until disease progression, unacceptable toxicity or patient's refusal.

The second- and subsequent lines of treatment will be at investigators' choice.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any study specific procedures. Subjects must be able to understand and willing to sign a written informed consent.
* Male or female subjects ≥ 18 years, expected lifespan ≥ 12 weeks.
* Patients have histologically or cytologically confirmed RAS and BRAF wild-type, MSS metastatic colorectal adenocarcinoma (mCRC), excluding appendiceal and anal cancers.
* AJCC/UICC stage IV left-side metastatic colorectal cancer. At least one measurable lesion according to RECIST 1.1.
* The patient has not previously received any systemic treatment specifically targeting advanced or metastatic colorectal cancer, including chemotherapy, monoclonal antibodies such as cetuximab or panitumumab targeting the epidermal growth factor receptor (EGFR), bevacizumab targeting the vascular endothelial growth factor (VEGF), immune checkpoint inhibitors such as anti-PD-1 or anti-PD-L1 antibodies, and anti-CTLA-4 antibodies. If recurrence or metastasis occurs during or within 6 months after adjuvant or neoadjuvant chemotherapy, adjuvant/neoadjuvant therapy is considered as a first-line systemic treatment for advanced or metastatic disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Within 7 days before treatment, the following laboratory test values are obtained and appropriate organ function is present:

Hemoglobin ≥ 90g/L, neutrophil count ≥ 1.5 × 10^9/L, platelet count ≥ 75 × 10^9/L; Serum total bilirubin ≤ 1.5 × upper limit of normal (UNL); Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 × UNL; if there are liver metastases, AST or ALT ≤ 5 × UNL; Serum creatinine ≤ 1.5 × UNL.

* Women of childbearing potential must have a negative blood pregnancy test at the baseline visit. For this trial, women of childbearing potential are defined as all women after puberty, unless they are postmenopausal for at least 12 continuous months, are surgically sterile, or are sexually inactive.
* Patients are not allowed to participate in other clinical trials during the study period and willing to comply with the study protocol and visit plan.

Exclusion Criteria:

* Concurrent active malignancy, excluding malignancies with disease-free survival of 5 years or more or in situ carcinoma considered cured after adequate treatment.
* Currently diagnosed with gastrointestinal diseases such as duodenal ulcer, ulcerative colitis, intestinal obstruction, or other conditions determined by the investigator to potentially cause gastrointestinal bleeding or perforation.
* Experienced thrombotic or embolic events, such as cerebrovascular accidents (including transient ischemic attacks), pulmonary embolism, or deep vein thrombosis, within the 12 months prior to study enrollment.
* Experienced the following conditions within the 12 months prior to study enrollment: myocardial infarction, severe/unstable angina pectoris, New York Heart Association (NYHA) class II or above heart failure, clinically significant supraventricular or ventricular arrhythmias, or symptomatic congestive heart failure.
* Use of systemic antibiotics for ≥7 days within the 4 weeks prior to study enrollment, or the occurrence of unexplained fever (>38.5°C) during the screening period/prior to the first dose (fever attributed to the tumor can be considered for enrollment, as determined by the investigator).
* Presence of uncontrolled pleural effusion, ascites, or pericardial effusion within 14 days prior to study enrollment despite appropriate treatment.
* Presence of any unresolved adverse events of Grade 2 or higher (excluding anemia, alopecia, and skin pigmentation) attributed to previous treatments according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
* Presence of interstitial lung disease, non-infectious pneumonia, or uncontrolled systemic diseases (e.g., diabetes, hypertension, pulmonary fibrosis, and acute pneumonia).
* Known human immunodeficiency virus (HIV) infection or known active hepatitis (defined as HBV-DNA ≥ 500 IU/ml for hepatitis B, and HCV-RNA above the limit of detection for hepatitis C) or co-infection with hepatitis B and C.
* History of known or suspected allergy to any investigational drug used in the study.
* Pregnancy or lactation in women.
* Pre-menopausal women (last menstrual period <2 years ago) who do not use or refuse to use effective non-hormonal contraception, or fertile men.
* Presence of other significant physical or mental illnesses or laboratory abnormalities that may increase the risk of participation in the study, interfere with study results, or are deemed unsuitable for participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2 year
  Time from date of randomization until the date of first documented progression or date of death from any cause, whichever came first.

SECONDARY OUTCOMES:
Objective response rate | 2 year
  CR + PR rate according to RECIST
Disease control rate | 2 year
  CR + PR + SD rate according to RECIST
No evidence of disease | 2 year
  The percentage of patients who had a curative treatment following protocol treatment, i.e., liver metastases that can be completely resected and/or ablated with no evidence of residual malignant disease.
Overall survival | 4 year
  Time from date of randomization until the date of first documented death from any cause.
Safety (Incidence of Adverse Events) | 2 year
  Percentage of patients, relative to the total of enrolled subjects, experiencing a specific adverse event of grade 3/4, according to National Cancer Institute Common Toxicity Criteria (version 5.0), during the induction and the maintenance phases of treatment.
Health related quality of life | Every 2 weeks after the first treatment until 6 months.
  Scores according to EORTC QLQ-CR29 scoring manual.
Quality-adjusted time without symptoms or toxicity | 2 year
  Q-TWiST was calculated as the sum of the utility-weighted mean durations for each health state. Q-TWiST = (TWiST × μTWiST) + (TOX × μTOX) + (REL × μREL).
  Base case utilities: μTWiST = 1, μTOX = 0.5, μREL = 0.5. Duration of AEs was measured until disease progression. All time in TOX was front-loaded at the beginning of threrapy.

OTHER OUTCOMES:
Tumor-infiltrating lymphocyte | 2 year
  Assessment of the tumor-infiltrating lymphocytes (TILs) in tumor tissue before treatment and during tumor progression.
Treatment-emergent genetic mutations (e.g., KRAS, NRAS, BRAF, SMAD4, HER2, Etc.) | 2 year
  Assessment of the correlation between mutation status of relevant genes and treatment response through ctDNA testing.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, Ph.D, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (3):
- China (3):
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Affiliated Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou